CLINICAL TRIAL: NCT05216822
Title: Role of Anti-Secretory Drug in Treatment of Children With Acute Watery Diarrhea
Brief Title: Anti-Secretory Drug in Treatment of Acute Watery Diarrhea
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam Roshdy Elkhayat, Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-2/2019AZA
Record Dates: First submitted 2021-12-06; First posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Acute Watery Diarrhea
MeSH Terms: interventions — racecadotril

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- children received ORS and racecadotril as treatment (Experimental): 25 children received ORS and racecadotril as treatment (at a dose of 1.5 mg/kg/day, an oral single daily dose for three days)
  Interventions: Drug: Racecadotril
- children received ORS alone as treatment (Active Comparator): 25 children received ORS alone for treatment as a control group
  Interventions: Drug: Racecadotril

INTERVENTIONS:
Drug: Racecadotril — racecadotril (dose of 1.5 mg/kg/day, an oral single daily dose for three days
  Other Names: Acetorphan

SUMMARY:
In conclusion, racecadotril is an anti-secretory drug that exerts its antidiarrheal effect by inhibiting intestinal enkephalinase. It is effective in reducing the volume and frequency of stool output. racecadotril is well tolerated and safe by providing symptomatic relief and reducing the severity of diarrhea as an adjuvant therapy during the acute attack of gastroenteritis. It is recommended that the new generations of already discovered drugs for control of secretory diarrhea should be studied to discover the ones with fewer side effects to other systems in the body.

DETAILED DESCRIPTION:
Background: Previous studies have shown that racecadotril is a safe and effective drug in treating children with acute diarrhea. Study Aim: to evaluate the effect of racecadotril as an adjunct to oral rehydration solution in the treatment of acute watery diarrhea among children under 5 years of age. Subjects and methods: This RCT trial included 50 children with acute watery diarrhea for 5 days or less with a frequency of three or more diarrheic stools in the past 24 hours before admission to the hospital, with no/mild to moderate dehydration.

ELIGIBILITY:
Inclusion Criteria:

* Age group for six months - 5 years.
* No or mild to moderate dehydration.
* Alert patient (to tolerate oral intake since the drug is only available in oral form).

Exclusion Criteria:

* Patients with severe dehydration (inability to drink because of drowsiness).
* Patients with any serious concomitant illness that needs antibiotic treatment.
* If severe adverse events occur at any time.
* Chronic diarrhea.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Diarrheal episode | 1-3 months
  number

CONTACTS AND LOCATIONS:
Overall Officials: Hamada M Kamel, MD, Principal Investigator — Professor
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No